CLINICAL TRIAL: NCT00584090
Title: Solifenacin Succinate (VESIcare) for the Treatment of Urinary Incontinence in Parkinson's Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn with intent of persuing larger, multi-site study.
Sponsor: University of South Florida (Other)
Responsible Party: Theresa Zesiewicz, MD, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4; 104803b
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2010-10

CONDITIONS: Urinary Incontinence; Parkinson's Disease
Keywords: urinary incontinence; parkinson's disease; vesicare; solifenacin succinate
MeSH Terms: conditions — Urinary Incontinence; Parkinson Disease | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Solifenacin Succinate (VESIcare)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solifenacin Succinate (VESIcare) — 5 - 10 mg po qd for 1 month
  Arms: 1
Drug: Placebo — Placebo equivalent of 5-10 mg po qd for 1 month
  Arms: 2

SUMMARY:
The primary purpose of this study is to measure the efficacy of solifenacin succinate (VESIcare) on treating urinary incontinence in Parkinson's disease patients.

The secondary objective of this study is to examine the effect of solifenacin succinate (VESIcare) on symptoms of PD and the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria.
2. Age 30 years to 80 years.
3. Stable dose of antiparkinsonian medication 4 weeks prior to study entry.
4. Patients must score 18 or higher on the UPDRS scale and 1.0 to 2.5 on the Modified Hoehn and Yahr scale.
5. Women of child-bearing potential must use a reliable method of contraception.
6. Must be experiencing symptoms of urinary incontinence (voiding 8 or more times/day or episodes of incontinence 5 or more times per week).
7. Patients must have evidence of normal PSA and urodynamic tests within the last 12 months.
8. Clearance from the patient's urologist or internist who has examined the patient within the last 12-months.

Exclusion Criteria:

1. Any illness that in the investigator's opinion preclude participation in this study.
2. Pregnancy or lactation.
3. Concurrent participation in another clinical study.
4. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam score less than 24).
5. Legal incapacity or limited legal capacity.
6. Presence of severe renal disease (BUN 50% greater than normal).
7. Presence of major hepatic impairment.
8. Currently taking ketaconazole (anti-fungal) or any CYP3A4 inhibitor.
9. Any history of bladder outflow obstruction or gastrointestinal obstructive disorders.
10. History of controlled narrow angle glaucoma.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
The primary purpose of this study is to measure the efficacy of solifenacin succinate (VESIcare) on treating urinary incontinence in Parkinson's disease patients. | 1 month

SECONDARY OUTCOMES:
The secondary objective of this study is to examine the effect of solifenacin succinate (VESIcare) on symptoms of PD and the patient's quality of life. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States